CLINICAL TRIAL: NCT00573846
Title: Phenotypic Characteristics of Inflammatory Bowel Disease in Southeast Asian Population - A Multi-centered US Study
Status: Withdrawn | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: University of Kentucky (Other); University of Texas Southwestern Medical Center (Other); Texas Health Resources (Other); Mayo Clinic (Other); Jefferson Medical College of Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Nimisha Parekh, Assistant Clinical Professor, University of California, Irvine
Other Study IDs: OCRT07005; 2007-5807
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective, case control study of inflammatory bowel disease. This study will analyze the phenotypic characteristics of inflammatory bowel disease in the Southeast Asian population and will help describe clinical characteristics and serologic profiles in Southeast Asians with inflammatory bowel disease, comparing the phenotype differences to historical Caucasian controls. The data from this study will help identify the phenotype characteristics of different ethnic groups and study the epidemiological patterns of the disease.

DETAILED DESCRIPTION:
This study is a retrospective, case control study of inflammatory bowel disease characteristics in patients with origins from the Indian sub-continent. Patients will be selected from the IBD registry maintained at respective institutions. Subjects from the Indian sub-continent will be identified using their country of birth, parents' ethnicity, number of years since leaving the country of birth, and number of years residing in the United States.

Using both electronic and paper databases, demographic information regarding age, gender, body mass index, smoking history, dietary habits; medical history such as type of IBD, IBD symptoms, location and behavior, medication use (past and current), history of other autoimmune disorders; surgical history (IBD and non-IBD related); laboratory indices such as IBD serology, Thiopurinemethyltransferase (TPMT), and infliximab levels will be collected.

Demographics will be compared between groups using descriptive statistics. Using univariate analysis, variables that are significantly different will be identified. Conditional logistic regression will then be performed to identify those clinical variables that are statistically significant.

The study duration will be one year from IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* Patients with origins from the Indian sub-continent
* Patients will be selected from the IBD registry maintained at respective institutions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected from the IBD registry maintained at respective institutions. Subjects from the Indian sub-continent will be identified using their country of birth, parents' ethnicity, number of years since leaving the country of birth, and number of years residing in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Phenotypic characteristics of inflammatory bowel disease in southeast asian population | 12 months
  Retrospective chart review

CONTACTS AND LOCATIONS:
Overall Officials: Nimisha K Parekh, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States